CLINICAL TRIAL: NCT04061759
Title: A Randomized Controlled Clinical Trial
Brief Title: Physiotherapy in Lumbar Disc Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guven Health Group (Other)
Responsible Party: Principal Investigator, GUL BALTACI, PROFESSOR, PT.PH.D., Guven Health Group
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 515
Record Dates: First submitted 2019-08-17; First posted 2019-08-20 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Lumbar Disc Disease; Lumbar Disc Herniation; Low Back Pain, Mechanical; Low Back Strain
MeSH Terms: conditions — Intervertebral disc disease; Intervertebral Disc Displacement; Low Back Pain | interventions — Reflexotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Soft tissue mobilization&stabilization exercises (Active Comparator): The following manual therapy techniques will be applied:
  1. Soft Tissue Mobilization;
  2. Pretzel Maneuvers;
  3. Pelvis Backward-Distraction;
  4. Trunk Rotation;
  5. Multifidus Mobilization; and
  6. Piriformis Transverse Friction Massage
  Interventions: Other: Effectiveness of four physical therapy approaches (soft tissue manual therapy, Kinesio® Taping techniques, stabilization exercises and reflex therapy) for treating lumbar disc pathologies.
- Kinesiotape&stabilization exercises (Active Comparator): The Kinesio® Taping muscle technique, with 10-25% of the stretch of the tape, will be applied to the sacrospinalis, quadratus lumborum, gluteus medius/maximus and piriformis muscles, based on the the weakness that patient's muscles had. Factors interfering with tape adhesion, such as sweat or hair, will be removed before the application. The tape can stay in place for 3-5 days due to its water resistant and breathable properties
  Interventions: Other: Effectiveness of four physical therapy approaches (soft tissue manual therapy, Kinesio® Taping techniques, stabilization exercises and reflex therapy) for treating lumbar disc pathologies.
- Stabilization exercises (Active Comparator): The core stabilization exercise treatment program consisted of the following exercises: a posterior pelvic tilt exercise, lower abdominal muscle isometric strengthening, hip adductor muscle isometric strengthening, lumbar stabilization exercises with a Swiss ball, upper and lower abdominal muscle strengthening exercises with a Swiss ball, oblique abdominal muscle strengthening exercises with a Swiss ball, quadratus lumborum muscle stretching with a Swiss ball, back extensor muscle strengthening exercises with a Swiss ball, a slump exercise (sciatic nerve stretching), lumbar lordosis exercises with a Swiss ball, bridge exercises with a Swiss ball, single leg bridge exercises on a Swiss ball, posture exercises, push-up exercises with a Swiss ball, and squat exercises with a Swiss ball
  Interventions: Other: Effectiveness of four physical therapy approaches (soft tissue manual therapy, Kinesio® Taping techniques, stabilization exercises and reflex therapy) for treating lumbar disc pathologies.
- Reflex therapy&Stabilization exercises (Active Comparator): Mobilization of each vertebra and pulls were applied from the medial side of the toe to the medial malleolus and to the heel by hand or with the help of an apparatus, including the cervical, thoracic and lumbar spine reflex zones. Finally, the procedure was finished by making a V-shaped maneuver with a thumb in the direction of spinal nerve exits.
  Interventions: Other: Effectiveness of four physical therapy approaches (soft tissue manual therapy, Kinesio® Taping techniques, stabilization exercises and reflex therapy) for treating lumbar disc pathologies.

INTERVENTIONS:
Other: Effectiveness of four physical therapy approaches (soft tissue manual therapy, Kinesio® Taping techniques, stabilization exercises and reflex therapy) for treating lumbar disc pathologies. — Visual analog scale (VAS) scores for pain intensity, goniometric measurements for the range of motion and hamstring flexibility, the sit and reach test for flexibility, an isokinetic evaluation for strength at 60°/sec, and a side-plank position test for trunk stabilization were measured. The functional status was evaluated with the Oswestry Disability Index. All groups were assessed at the beginning, after a four-week treatment and four weeks of follow-up.

SUMMARY:
The aim of this study is to compare the effectiveness of four physical therapy treatment approaches for lumbar region pathologies. Eighty volunteers who have back pain will be included in the study. Subjects will be randomly divided into four groups; Group 1: Soft tissue mobilisation techniques and stabilization exercises (n=20), Group 2: Kinesiotape and stabilization exercise (n=20), Group 3: Stabilization exercises (n=20), Group 4: Reflexology and stabilization exercises (n=20).

DETAILED DESCRIPTION:
All patients will be measured with visual analog scale for pain level, goniometric measurement for range of motion, hamstring tension and sit and reach for flexibility, isokinetic evaluation for strength in 60degree/ sec, Side plank position test for trunk stabilization.

Function will be measured with Oswestry Disability Index. Manual muscle testing for flexion, extension, lateral flexion of back, flexion, extension, abduction of hip, flexion, extension of knee and inversion, eversion of ankle will be assessed. Group 1, 2 and 4 will be started to treatment twice a week for 4 weeks after first evaluation. Group 3 will be had home exercise programme after first evaluation.

Groups will be assessed again at 4th and 8th weeks after treatment. Multiway variant analysis will bee done within each group before the treatment and at follow-up. When differences observed, Tukey test will be used to find out the group that caused the differences.

ELIGIBILITY:
Inclusion Criteria:

* The participants between the ages of 25 and 55 years,
* Having a minimum pain level (at activity) of 3 out of 10 on visual analog scale
* Having low back pain for at least 3 months with lumbar disc pathology (bulging or protrusion) diagnosed by clinical tests and magnetic resonance imaging.

Exclusion criteria:

* sacroiliac and lumbar degenerative pathologies,
* another pathology related to neurological deficits,
* physiotherapy previously received for at least 12 months,
* any surgery affecting the lumbar region.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
pain intensity | 8weeks
  All patients will be assessed with the visual analog scale (VAS) for pain intensity at rest, at night and during activity. VAS is a 100-mm line with no marks along it, anchored with the words "no pain" on one side and "the most severe pain" on the other. The subjects were simply instructed to place a mark along the line at a level representing the intensity of their pain.
range of motion | 8weeks
  Trunk and hip range of motion measurements were taken with a universal goniometer. Active trunk flexion and extension, lateral flexion, and hip flexion and extension will recorded. Hamstring flexibility will be also measured with universal goniometry using the passive 90/90 test. For this test, the patients will be positioned supine, lying on the back, with the knee and hip stabilized at 90° of flexion. The goniometer will be pivoted at the lateral condyle of the femur, and knee extension will be measured in order to determine the loss of the range of motion due to hamstring tightness.
muscular strength | 8weeks
  All patients were assessed with isokinetic testing for strength at 60°/sec. Isokinetic testing is commonly used for testing and training of patients in clinics. It calculates the muscle power at the full range of motion, providing the opportunity to act at the angular velocity. An IsoMed 2000 (D&R GmbH, Germany) will be used bilaterally for isokinetic evaluation of hip flexion and abduction at 60°/sec. After proper positioning, the patient will be asked to push the force arm of the system as strongly as possible at this angular velocity in the flexion and abduction directions. The peak torque and total work values will be recorded.
Trunk stabilization test | 8weeks
  A side-plank position test was used for evaluation of trunk stabilization. The test is one of the most functional stabilization tests and examines trunk strength, endurance and stabilization during synchronized extremity movements. Basically, the lateral core muscles are assessed but oblique abdominal muscles and hip flexors are also examined. Patients are positioned in side lying, with 90° elbow flexion, 60° shoulder abduction, legs extended and whole body aligned. After trial repetition, patients are asked to raise their pelvis off the ground and stay in that position as long as possible without disrupting the smoothness of the motion. The test is finished when the position is disrupted or the patient falls.
Functional performance | 1hour
  The functional status will be evaluated with the Oswestry Disability Index. Knowing the symptoms and disabilities of low back pain patients gives us valuable information for planning the treatment process. The Oswestry Disability Index has 10 main topics, namely, pain intensity, self-care, lifting, walking, sitting, standing, sleep quality, sexual function, social life, and traveling. Each section is scored from 0 to 5 points. The degree of disability increases as the score increases.

CONTACTS AND LOCATIONS:
Overall Officials: Yesim Sardan Cetinkaya, MD, Study Director — Guven Health Group
Locations (1):
- Anima Rapha Center, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Standaert CJ, Weinstein SM, Rumpeltes J. Evidence-informed management of chronic low back pain with lumbar stabilization exercises. Spine J. 2008 Jan-Feb;8(1):114-20. doi: 10.1016/j.spinee.2007.10.015. PMID 18164459
- [Result] Burns SA, Cleland JA, Rivett DA, Snodgrass SJ. Effectiveness of physical therapy interventions for low back pain targeting the low back only or low back plus hips: a randomized controlled trial protocol. Braz J Phys Ther. 2018 Sep-Oct;22(5):424-430. doi: 10.1016/j.bjpt.2018.08.014. Epub 2018 Sep 7. PMID 30217693
- [Result] Burns SA, Cleland JA, Cook CE, Bade M, Rivett DA, Snodgrass S. Variables Describing Individuals With Improved Pain and Function With a Primary Complaint of Low Back Pain: A Secondary Analysis. J Manipulative Physiol Ther. 2018 Jul-Aug;41(6):467-474. doi: 10.1016/j.jmpt.2017.11.006. Epub 2018 Aug 9. PMID 30100096
- See also: related physiotherapy techniques for lumbar spine pathology — http://www.spine-health.com